CLINICAL TRIAL: NCT04027855
Title: A Study on the Collection of Peripheral Blood Mononuclear Cells From Healthy Volunteers for the Development of Allogeneic Cellular Immunotherapy Products
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Both the sponsors and collaborator are considering terminating the study
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Legend Biotechnology Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, WEI XU, Chief Physician of hematology department, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BM2L201903
Record Dates: First submitted 2019-07-19; First posted 2019-07-22 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Collection of Peripheral Blood Mononuclear Cells by Means of Apheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collection of PBMC from healthy donors (Other): 1. Screening period: All volunteers are required to sign a written informed consent form for the study; after the signing of informed consent form, the demographic data and medical history of the volunteers will be collected, and physical examinations and local laboratory tests will be performed to assess the eligibility of the volunteers. Volunteers who meet all the inclusion criteria and do not meet any exclusion criteria (except for the basic biological indicators of UCAR-T product preparation) will receive peripheral venous whole blood sampling, and the volunteers receiving apheresis based on the assessment results will be enrolled.
  2. Apheresis period: 5 volunteers who meet the inclusion criteria will undergo collection of peripheral blood mononuclear cells (PBMC) by means of apheresis.
  Interventions: Procedure: collection of peripheral blood mononuclear cells from healthy volunteers

INTERVENTIONS:
Procedure: collection of peripheral blood mononuclear cells from healthy volunteers — 1. Screening period: All volunteers are required to sign a written informed consent form for the study; after the signing of informed consent form, the demographic data and medical history of the volunteers will be collected, and physical examinations and local laboratory tests will be performed to assess the eligibility of the volunteers. Volunteers who meet all the inclusion criteria and do not meet any exclusion criteria (except for the basic biological indicators of UCAR-T product preparation) will receive peripheral venous whole blood sampling, and the volunteers receiving apheresis based on the assessment results will be enrolled.
  2. Apheresis period: 5 volunteers who meet the inclusion criteria will undergo collection of peripheral blood mononuclear cells (PBMC) by means of apheresis.

SUMMARY:
The objective of the study is to collect peripheral blood mononuclear cells (PBMC) from healthy volunteers for the research and development of allogeneic cellular immunotherapy products.

DETAILED DESCRIPTION:
The study is a single-center study.

1. Screening period: All volunteers are required to sign a written informed consent form for the study; after the signing of informed consent form, the demographic data and medical history of the volunteers will be collected, and physical examinations and local laboratory tests will be performed to assess the eligibility of the volunteers. Volunteers who meet all the inclusion criteria and do not meet any exclusion criteria (except for the basic biological indicators of UCAR-T product preparation) will receive peripheral venous whole blood sampling, and the volunteers receiving apheresis based on the assessment results will be enrolled.
2. Apheresis period: 5 volunteers who meet the inclusion criteria will undergo collection of peripheral blood mononuclear cells (PBMC) by means of apheresis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 40 years, male or female;
2. Weight: male ≥ 50 kg, female ≥ 45 kg; 18.5 ≤ BMI ≤ 30;
3. Healthy volunteers who signed informed consent form.

Exclusion Criteria:

1. Those with known respiratory, circulatory, digestive, urinary, blood, immune, endocrine disorders or metabolic disorders;
2. Those with known neurological diseases, mental illnesses, Creutzfeldt-Jakob disease and those with a family history, or those treated with tissue or tissue derivatives that may be derived from Creutzfeldt-Jakob infected people;
3. Those with known chronic skin diseases, especially infectious, allergic or inflammatory systemic skin diseases;
4. Those with known allergic diseases or recurrent allergies;
5. Those with known malignant tumors or health-affecting benign tumors;
6. Two or more physical examination results of blood pressure have shown (except for white coat hypertension): systolic blood pressure < 90 or ≥ 140mmHg, or diastolic blood pressure < 60 or ≥ 90 mmHg, or pulse pressure difference < 30 mmHg, heart rate: < 60 beats/min or >100 beats/min;
7. Laboratory tests: hemoglobin determination: male <120 g/L, female <115 g/L, or liver and kidney function is more than 1.5 times the upper limit of normal and clinically significant, or 12-lead ECG is abnormal and clinically significant, or abdominal B-mode ultrasound is abnormal and clinically significant, or chest X-ray is abnormal and clinically significant, and T cell detection of tuberculosis infection is over the limit or positive;
8. lymphocyte subsets （lymphocyte proportion、CD3+、CD3+CD4+、CD3+CD8+、CD3-CD16+CD56+、CD19+）Abnormal detection and clinical significance;
9. Those with positive hepatitis B surface antigen or HBV DNA, or hepatitis B e antigen, or hepatitis C antibody, or Treponema pallidum antibody, or human immunodeficiency virus antibody;
10. Recipients of allogeneic tissue and organ transplants;
11. Those who have undergone resection of vital internal organs such as stomach, kidney, spleen and lung;
12. Those who have suffered from blood transfusion-associated infectious diseases;
13. Those who have undergone minor surgery within less than 3 months, such as appendectomy and ophthalmic surgery; those who have undergone major surgery within less than 1 year, such as surgical treatment for gynecological benign tumors or superficial benign tumors;
14. Women who are pregnant, or have an abortion within less than 6 months or have undergone less than 1 year after childbirth and lactation;
15. Those whose upper respiratory tract infection has recovered for less than 1 week, or pneumonia has recovered for less than 3 months;
16. Those whose acute pyelonephritis has recovered for less than 3 months, or those with acute exacerbation of urinary calculi;
17. Those who have been injured or wound-contaminated by equipment contaminated by blood or tissue fluids, or who have got a tattoo for less than 1 year;
18. Those who have received whole blood and blood component transfusion within 1 year;
19. Those who have received the last vaccination of live attenuated vaccines such as measles, mumps, or polio within 2 weeks, or have received the last vaccination of rubella live vaccine, human rabies vaccine, live attenuated Japanese encephalitis vaccine within 4 weeks;
20. Those who have received the last vaccination of rabies vaccines after being bitten by an animal within 1 year;
21. Those who have received the last vaccination of antitoxin or immune serum injection within 4 weeks, or those who have received the last vaccination of hepatitis B human immunoglobulin injection within 1 year;
22. Those who have participated in clinical trials within 1 month; if they have used investigational drugs, they need to be discussed case by case;
23. Those who cannot meet the basic biological indicators for UCAR-T product preparation, specifically including positive blood safety indicator sterility test result, or positive mycoplasma test result, or culture product endotoxin test ≥ 10 EU/mL; basic biological indicator cell viability is < 70%, or the number of effective T lymphocytes cannot meet the needs of in vitro assessment, or the in vitro proliferative production characteristics of each component cell, or the proportion of each component cannot meet the UCAR-T preparation conditions;
24. Those who are considered by the investigator as unsuitable for participating in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
the number of PBMC | two year

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, PhD& MD, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China